CLINICAL TRIAL: NCT02175485
Title: Evaluation of Efficacy of Dellegra® Combination Tablet (Fexofenadine Hydrochloride 30mg /Pseudoephedrine Hydrochloride 60mg) in Allergic Rhinitis After Japanese Cedar Antigen Exposure in Japanese Population. Open Label Study
Brief Title: Evaluation of Efficacy of Dellegra in Exposure Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEXHYL06934; U1111-1152-0373 (Other: UTN)
Record Dates: First submitted 2014-06-22; First posted 2014-06-26 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fexofenadine HCl (Experimental): 2 tablets of Dellegra Combination Tablets (Fexofenadine Hydrochloride 30 mg+Pseudoephedrine Hydrochloride 60 mg/tablet), oral, administrated 2 hours after start of exposure with 8,000 grains/cubic meter of Japanese cedar pollen
  Interventions: Drug: Fexofenadine HCl 30 mg+Pseudophedrine HCl 60 mg

INTERVENTIONS:
Drug: Fexofenadine HCl 30 mg+Pseudophedrine HCl 60 mg — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To collect and analyze clinical data of Allergic Rhinitis patients' Total Nasal Symptom Score (TNSS) change after Dellegra internal use under high density pure Japanese cedar pollen exposure.

Secondary Objective:

To collect and analyze clinical data of Allergic Rhinitis patients' change in Total Symptom Score (TSS) and amount of nasal discharge, safety, and overall patients' impression about efficacy of Dellegra after Dellegra internal use under high density pure Japanese cedar pollen exposure.

DETAILED DESCRIPTION:
It will be 8 days at minimum and up to 17 days depending on screening visit and post-treatment observation allowances.

ELIGIBILITY:
Inclusion criteria:

* Patients with seasonal allergic rhinitis.
* Patients with a history of symptoms of Japanese cedar pollinosis for at least 2 years.
* Positive radioallergosorbent test (RAST) for Japanese cedar pollen antigen (CAP-RAST class >=2) within 1.5 years before the exposure test.
* Patients with Total Nasal Symptom Score of 8 or more, and nasal congestion scores of 2 (moderate) or more at least 1 assessment point of 90 to 150 minutes after the start of the screening exposure.
* Age ≥20 and ≤65 years.
* Patients written informed consent.

Exclusion criteria:

* Patients with symptoms of perennial allergic rhinitis.
* Patients with severe asthma, bronchiectasis, severe hepatic, renal, or cardiac dysfunction, hematological, endocrine disease, and other serious complications.
* Patients with nasal diseases (hypertrophic rhinitis, paranasal sinusitis, nasal polyps, deviation of the nasal septum, etc.) or eye diseases that could interfere with judgment of the efficacy of Dellegra Combination Tablets.
* Patients with evidence of upper and/or lower respiratory tract inflammation (acute rhinitis, chronic rhinitis, congestive rhinitis, atrophic rhinitis, purulent nasal discharge, sinusitis in the presence of cold-like, etc.) on the day of treatment exposure.
* Patients who have taken any of the following medications that may affect the evaluation of Dellegra Combination Tablets (except for the use of topical preparation in which investigator/sub-investigator judged them not to affect the efficacy evaluation; the treated site is different, etc.):
* Within 2 weeks prior to the day of the screening exposure test: Antiallergic drugs, antihistamines (H1 and H2 blockers: oral administration, nose drops, eye drops, injection, and topical use), anticholinergic agents, vasoconstrictor nose drops, antihistamine-containing cold remedies, agents that can be expected to have an antiallergic/antihistaminic effect (including Chinese medicines and glycyrrhizin), and other agents that are indicated for allergic symptoms (sneezing, rhinorrhea, nasal congestion, and eye itching etc.). Steroids (oral, inhaled, nose drops, eye drops, or topical use), immunosuppressants (oral, topical use, or injected), azole fungicides, and histamine containing gamma-globulin preparations.
* Within 4 weeks prior to the day of the screening exposure test: Depot steroid preparations.
* Patients who are considered by the investigator/sub-investigator to be unsuitable for enrollment in the study for any other criterion.
* Patients with a history of hypersensitivity to antihistamines or antihistaminic agent (fexofenadine HCI is included), and the pseudoephedrine hydrochloride.
* Patients with severe hypertension or severe coronary artery disease, narrow angle glaucoma, urinary retention, or those who have shown sensitivity to adrenergic agents (manifestations include insomnia, dizziness, weakness, tremor, or arrhythmias).
* Women who are pregnant, may be pregnant, or currently breast-feeding.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean change in Total Nasal Symptom Score (sneezing, nasal discharge, nasal congestion, and itchy nose | From 2 hours after antigen exposure (baseline) to 3 hours after intake of Dellegra

SECONDARY OUTCOMES:
Mean change of Total Symptom Score (sneezing, nasal discharge, nasal congestion, itchy nose, lacrimation, and eye itching | Prior to exposure, and every 15 minutes for 5 hours after exposure start
Overall patients' impression about efficacy of Dellegra after Dellegra internal use (Score 1 [none] to 7 [very severe]) | From intake of Dellegra up to 17 days
Number of patients who experienced adverse events | From intake of Dellegra up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392-001, Shinjuku-ku, Japan